CLINICAL TRIAL: NCT04246879
Title: Diagnostic Accuracy of Delayed MRI Contrast Enhancement Characteristics and Radiation Necrosis Following Stereotactic Radiosurgery (SRS) for Brain Metastases
Brief Title: MRI Following Stereotactic Radiosurgery (SRS) for Brain Metastases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00103163
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
Keywords: Laser Interstitial Thermal Therapy (LITT); Stereotactic radiosurgery (SRS); Magnetic resonance image (MRI)
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Experimental)
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Subjects undergo one additional delayed MRI sequence

SUMMARY:
The purpose of this study is to test whether an additional magnetic resonance image (MRI) sequence can improve the ability to distinguish radiation damage from tumor recurrence in participants with brain metastasis who have previously been treated with stereotactic radiosurgery (SRS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥18
* Metastatic malignancy with at least 1 brain metastasis previously treated with SRS
* Patients may have also received whole brain radiation therapy (WBRT) for management of brain metastatic disease but this is not required for study participation
* Patients must have been diagnosed with a metastatic solid tumor of any histological type except small cell lung cancer (SCLC), or lymphoma.
* Radiographic progression on post-SRS imaging at previously treated SRS site(s)
* Must be a candidate for brain surgery as determined by treating neurosurgeon and/or anesthesia team
* Patients must sign study-specific informed consent prior to study entry

Exclusion Criteria:

* Poor surgical candidate as determined by treating neurosurgeon and/or anesthesia team
* Unable to undergo contrasted MRI (e.g. incompatible medical device, inadequate renal function per standard institutional clinical protocol, contrast allergy)
* Small cell lung cancer (SCLC) or lymphoma histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
number of positive MRI sequences along with positive tumor biopsies | baseline
  true tumor will be detected by delayed MRI as determined by biopsy
number of negative MRI sequences along with negative tumor biopsies | baseline
  absence of tumor will be detected by delayed MRI as determined by biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Scott Floyd, M.D. Ph.D., Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No